CLINICAL TRIAL: NCT01819038
Title: Early Renal Replacement Therapy and the Outcome of Acute Kidney Injury
Acronym: EarlyRRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Principle Investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: chula
Record Dates: First submitted 2013-03-18; First posted 2013-03-27 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-12

CONDITIONS: Acute Renal Failure
MeSH Terms: conditions — Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High NGAL and early RRT (Experimental): NGAL level > 400 ng/ml and start continuous renal replacement therapy early
  Interventions: Procedure: continuous renal replacement therapy
- High NGAL and late RRT (Experimental): NGAL > 400 ng/ml and start continuous renal replacement therapy late
  Interventions: Procedure: continuous renal replacement therapy
- Low NGAL (Active Comparator): NGAL < 400 ng/ml and starting continuous renal replacement therapy follow with absolute indication
  Interventions: Procedure: continuous renal replacement therapy

INTERVENTIONS:
Procedure: continuous renal replacement therapy

SUMMARY:
This research project is a prospective study to compare mortality between early renal replacement therapy (RRT) and late renal replacement therapy by using plasma neutrophil gelatinase associated lipocalin (pNGAL) as a tool in decision- making.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* patients with acute kidney injury in the intensive care ward.

Exclusion Criteria:

* The patient refuses to sign the consent
* The patient is pregnant, parturient, or breastfeeding
* End stage renal disease
* Chronic renal failure
* previous kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
mortality rate | 28 day

SECONDARY OUTCOMES:
ventilator free-days | 28 days

OTHER OUTCOMES:
hemodialysis free-days | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Nattachai Srisawat, M.D., Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787